CLINICAL TRIAL: NCT00327444
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-arm Study of the Effect of Intravenous Aflibercept Administered Every 2 Weeks in Advanced Ovarian Cancer Patients With Recurrent Symptomatic Malignant Ascites
Brief Title: Study of the Effect of Intravenous AVE0005 (VEGF Trap) in Advanced Ovarian Cancer Patients With Recurrent Symptomatic Malignant Ascites
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC6125; EudraCT : 2005-005026-31; AVE0005A /3001
Record Dates: First submitted 2006-05-16; First posted 2006-05-18 (Estimated); Results first posted 2013-01-01 (Estimated); Last update posted 2013-01-01 (Estimated); Status verified 2011-07

CONDITIONS: Ovarian Neoplasms; Ascites
Keywords: Ovarian neoplasm; Ascites; Angiogenesis inhibitor; Vascular Endothelial Growth Factor A; Recombinant fusion protein
MeSH Terms: conditions — Ovarian Neoplasms; Ascites | interventions — aflibercept

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Participants with advanced ovarian cancer administered placebo in the double-blind (DB) period.
  In the open-label (OL) period, participants had the option to receive aflibercept or be withdrawn from the study.
  Interventions: Drug: Placebo; Drug: aflibercept (ziv-aflibercept, AVE0005, VEGF trap, ZALTRAP®)
- Aflibercept (Experimental): Participants with advanced ovarian cancer administered aflibercept in the double-blind (DB) period.
  In the open-label (OL) period, participants had the option to continue to receive aflibercept or be withdrawn from the study.
  Interventions: Drug: aflibercept (ziv-aflibercept, AVE0005, VEGF trap, ZALTRAP®)

INTERVENTIONS:
Drug: aflibercept (ziv-aflibercept, AVE0005, VEGF trap, ZALTRAP®) — 4.0 mg/kg aflibercept was administered intravenously (IV) over 1 hour once every 2 weeks in the DB period.
  Arms: Aflibercept
Drug: Placebo — Placebo was administered intravenously (IV) over 1 hour once every 2 weeks in the DB period.
  Arms: Placebo
Drug: aflibercept (ziv-aflibercept, AVE0005, VEGF trap, ZALTRAP®) — 4.0 mg/kg aflibercept was administered intravenously (IV) over 1 hour once every 2 weeks in the OL period.

SUMMARY:
This study was designed to characterize the effect of aflibercept in participants with advanced chemoresistant ovarian cancer.

Primary objective: Compare the effect of aflibercept (ziv-aflibercept, AVE0005, VEGF trap, ZALTRAP®) to placebo treatment on repeat paracentesis in symptomatic malignant ascites in participants with advanced ovarian cancer

Secondary objectives: Safety, tolerability, paracentesis-related parameters, participant-reported outcome.

DETAILED DESCRIPTION:
The study included:

* A Thirty (30)-day screening phase
* The double blind treatment period for a minimum of 60 days. Day 1 of the double-blind treatment period was defined as the date of the qualifying paracentesis (ie, withdrawal of >= 1 Liter of ascitic fluid). Participants were randomized after adequate recovery from the qualifying paracentesis (The first dose was administered on Day 1 or Day 2).
* The optional open-label extension (until treatment discontinuation criteria were met)
* A posttreatment follow-up phase lasting 60 days.

Criteria for discontinuation included:

1. Participant or his legally authorized representative request discontinuation
2. In the Investigator's opinion, continuation of treatment would be detrimental to the participant's well being, such as disease progression, unacceptable toxicity, noncompliance, or logistical considerations
3. Sponsor request
4. Intercurrent illness that prevented further administration of investigational product(IP)
5. More than 2 IP dose reductions
6. Unacceptable adverse events (AE) not manageable by symptomatic therapy, dose delay, or dose modification
7. Arterial thromboembolic events, including cerebrovascular accidents, myocardial infarctions, transient ischemic attacks, new onset or worsening of preexisting angina
8. Radiographic evidence of intestinal obstruction (for example, dilated loops of bowel accompanied by air-fluid levels) or gastrointestinal perforation (for example, presence of extraluminal gas) requiring surgical intervention

ELIGIBILITY:
Participants who met the following criteria were eligible to participate in this study.

Inclusion Criteria:

* Advanced ovarian epithelial cancer, treated with paracentesis
* Platinum-resistant, and topotecan-resistant and/or liposomal doxorubicin-resistant disease;
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2.

Exclusion Criteria:

* Pseudomyxoma peritonei or peritoneal mesothelioma;
* Transudative ascites;
* Peritoneovenous or other shunt placed for malignant ascites management;
* Recent (<6 months) cardiovascular event (pulmonary embolus, myocardial infarction, stroke) or gastrointestinal disease (ulcer, hepatic cirrhosis);
* Known brain metastases;
* Uncontrolled hypertension;
* Recent treatment with chemotherapy, surgery or radiotherapy;
* Prior treatment with VEGF or VEGFR inhibitor.

The above information is not intended to contain all considerations relevant to participation in a clinical trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2006-07; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Walter GOTLIEB, Principal Investigator — Director of Gynecologic Oncology and Colposcopy Associate Professor of Oncology, McGill University - Montreal - Quebec Canada
Locations (9):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Vienna, Austria
- Sanofi-Aventis Administrative Office, Diegem, Belgium
- Sanofi-Aventis Administrative Office, Laval, Canada
- Sanofi-Aventis Administrative Office, Budapest, Hungary
- Sanofi-Aventis Administrative Office, Mumbai, India
- Sanofi-Aventis Administrative Office, Netanya, Israel
- Sanofi-Aventis Administrative Office, Barcelona, Spain
- Sanofi-Aventis Administrative Office, Guildford Surrey, United Kingdom

REFERENCES:
- [Derived] Gaitskell K, Rogozinska E, Platt S, Chen Y, Abd El Aziz M, Tattersall A, Morrison J. Angiogenesis inhibitors for the treatment of epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD007930. doi: 10.1002/14651858.CD007930.pub3. PMID 37185961
- [Derived] Gotlieb WH, Amant F, Advani S, Goswami C, Hirte H, Provencher D, Somani N, Yamada SD, Tamby JF, Vergote I. Intravenous aflibercept for treatment of recurrent symptomatic malignant ascites in patients with advanced ovarian cancer: a phase 2, randomised, double-blind, placebo-controlled study. Lancet Oncol. 2012 Feb;13(2):154-62. doi: 10.1016/S1470-2045(11)70338-2. Epub 2011 Dec 20. PMID 22192729

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Fifty-eight (58) participants from a total of 23 sites in 7 countries were enrolled in the study.
Pre-assignment Details: 55 were randomized (started population). 3 participants were not randomized but they were treated, and permanently withdrawn from the study due to disease progression (1 participant), fatal disease progression (1 participant) and a treatment emergent adverse event (1 participant).
Groups:
- Placebo: Participants with advanced ovarian cancer administered placebo intravenously, once every two weeks in the DB period and 4.0 mg/kg aflibercept intravenously, once every two weeks in the OL period.
- Aflibercept: Participants with advanced ovarian cancer administered 4.0 mg/kg aflibercept intravenously, once every two weeks in the DB period and the OL period.
Period: Double Blind Treatment (DB) Period
Arm/Group | Placebo | Aflibercept
Started | 26 | 29
SAFETY | 25 (Excludes one participant from the Placebo arm who received aflibercept in error in the DB period.) | 30 (Includes 1 from Placebo who received aflibercept in DB period)
Completed | 0 | 0
Not Completed | 26 | 29
Not completed — Disease progression | 10 | 13
Not completed — Adverse Event | 5 | 5
Not completed — Subject request | 0 | 1
Not completed — Withdrew DB and continued to OL | 11 | 10
Period: Open Label Treatment (OL) Period
Arm/Group | Placebo | Aflibercept
Started | 11 | 10
ONGOING TREATMENT | 1 | 0
Completed | 0 (All participants were treated till they met treatment discontinuation criteria) | 0 (All participants were treated till they met treatment discontinuation criteria)
Not Completed | 11 | 10
Not completed — Disease progression | 8 | 7
Not completed — Adverse Event | 2 | 2
Not completed — Worsening dyspnea | 0 | 1
Not completed — Ongoing Treatment | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Aflibercept | Total
Number analyzed (Participants) | 26 | 29 | 55
Age, Customized [Number; unit: participants] — Baseline characteristics are reported for the randomized population
  participants
    < 35 years | 0 | 1 | 1
    >=35 to <45 years | 5 | 1 | 6
    >=45 to <55 years | 10 | 7 | 17
    >=55 to <65 years | 4 | 11 | 15
    >=65 to <75 years | 6 | 7 | 13
    >=75 years | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 29 | 55
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 19 | 22 | 41
  Black | 1 | 0 | 1
  Asian, Oriental | 6 | 7 | 13

OUTCOME MEASURES:

1. Primary Outcome: Time to Repeat Paracentesis (TRP)
Description: TRP was defined as the number of days between the date of randomization and the date of the first post-randomization paracentesis.
  For participants who did not undergo a postrandomization paracentesis on study, TRP was calculated from randomization to the end of the double-blind treatment period.
Time Frame: From Day 1 up to 6 months from randomization
Population: The intent-to-treat (ITT) population - all participants who were randomized in the study.
Measure: Least Squares Mean (Standard Error); unit: days
Arm/Group | Placebo | Aflibercept
Number analyzed (Participants) | 26 | 29
days | 23.3 (7.70) | 55.1 (7.25)
Statistical Analysis 1: Comparison: Placebo vs Aflibercept; Test type: Superiority or Other; p = 0.0019, ANOVA — Estimated using Wilcoxon rank-sum test with stratification of baseline paracentesis (=<2 weeks versus >2 weeks) at randomization; Estimated from ANOVA model with stratification of baseline paracentesis (=<2 weeks versus >2 weeks); Least squares (LS) Mean difference = 31.8, 95% CI 2-sided [10.56 to 53.05], Standard Error of Mean 10.59 — The LS mean difference is estimated for aflibercept versus placebo (aflibercept-placebo)

2. Secondary Outcome: Area Under the Curve (AUC) for Participant Assessed Ascites Impact Measure (AIM)
Description: AIM 4 symptoms (abdominal discomfort, abdominal bloating, abdominal pain, and ability to move normally) are scored from 0 to 5, where higher scores represent worst outcomes. An AIM total score ranges from 0-20.
  A plot for (The AIM questionnaire total score - Baseline score) versus time were generated. AIM AUC represents the overall improvement (scored positive) if the area is below the baseline value or worsening (scored negative) if the area is above the baseline. AIM AUC for a participant is the sum of individual areas representing improvement (+) or worsening (-).
Time Frame: From Day 1 up to 60 days from randomization to the first postrandomization paracentesis
Population: The intent-to-treat (ITT) population - all participants who were randomized in the study, and had evaluable AIM scores.
Measure: Least Squares Mean (Standard Error); unit: (units on a 4-symptom scale)*day
Arm/Group | Placebo | Aflibercept
Number analyzed (Participants) | 15 | 16
(units on a 4-symptom scale)*day | 29.8 (148.07) | 405.3 (143.21)
Statistical Analysis 1: Comparison: Placebo vs Aflibercept; Test type: Superiority or Other; p = 0.0160, ANOVA — [p-value comment as in outcome 1, analysis 1]; Estimated from ANOVA model with stratification of baseline paracentesis (=<2 weeks versus >2 weeks); Least squares (LS) Mean difference = 375.5, 95% CI 2-sided [-46.48 to 797.42], Standard Error of Mean 205.99 — The LS mean difference was estimated for aflibercept versus placebo (aflibercept-placebo)

3. Secondary Outcome: 60-Day Frequency of Paracentesis (FOP)
Description: 60-Day FOP was defined as the total number of paracenteses performed within the first 60 days after randomization during the double blind treatment period.
Time Frame: From Day 1 up to 60 days from randomization
Population: The intent-to-treat (ITT) population - all participants who were randomized in the study.
Measure: Least Squares Mean (Standard Error); unit: paracentesis
Arm/Group | Placebo | Aflibercept
Number analyzed (Participants) | 26 | 29
paracentesis | 5.1 (0.69) | 2.7 (0.65)
Statistical Analysis 1: Comparison: Placebo vs Aflibercept; Test type: Superiority or Other; p = 0.0035, ANOVA — [p-value comment as in outcome 1, analysis 1]; Estimated from ANOVA model with stratification of baseline paracentesis (=<2 weeks versus >2 weeks); Least squares (LS) Mean difference = -2.4, 95% CI 2-sided [-4.33 to -0.54], Standard Error of Mean 0.94 — The LS mean difference is estimated for aflibercept versus placebo (aflibercept-placebo)

4. Secondary Outcome: Plasma Levels of Free and VEGF-bound Aflibercept
Description: Free aflibercept and VEGF-bound aflibercept plasma concentrations were measured by separate enzyme-linked immunosorbent assay (ELISA). The limit of quantitation of free aflibercept was 15.6 ng/mL, and of VEGF-bound aflibercept was 43.9 ng/mL.
  Peak free aflibercept was estimated at the end of Cycle 1 (C1) administration. The median free and VEGF-bound trough concentrations were determined for each participant beyond Cycle 3 (C3), then mean values were estimated from these median values.
Time Frame: Following every biweekly treatment administration up to 60 days after treatment discontinuation
Population: The analysis was performed using the safety population with evaluable blood samples. 42 participants were evaluated.
Measure: Mean (Standard Deviation); unit: μg/mL
Groups:
- Double Blind (DB) Period: Participants with advanced ovarian cancer administered placebo or 4.0 mg/kg aflibercept intravenously, once every two weeks in the DB period.
- Open-Label (OL) Period: Participants with advanced ovarian cancer administered 4.0 mg/kg aflibercept intravenously, once every two weeks in the OL period.
Arm/Group | Double Blind (DB) Period | Open-Label (OL) Period
Number analyzed (Participants) | 30 | 21
μg/mL
  Peak Free Aflibercept (C1) (N=20, N=15) | 69.8 (29.7) | 62.1 (29.5)
  Trough Free Aflibercept (Beyond C3) (N=15, N=19) | 5.33 (3.67) | 5.10 (5.29)
  Trough Bound Aflibercept (Beyond C3) (N=16, N=17) | 3.02 (1.29) | 3.49 (1.48)

ADVERSE EVENTS:
Time Frame: From treatment initiation to October 30, 2009
Description: Adverse events were collected and reported per arm only as there was no washout period between the double-blind and open label treatment periods.
Arm/Group | Placebo | Aflibercept
Serious Adverse Events (participants affected / at risk) | 18/25 | 27/30
Other Adverse Events (participants affected / at risk) | 22/25 | 28/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=25) | Aflibercept (N=30)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 3
Ascites (Gastrointestinal disorders) | 2 | 1
Colonic fistula (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 2 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 2
Obstruction gastric (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 3
Small intestinal perforation (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 6
Asthenia (General disorders) | 0 | 1
Death (General disorders) | 0 | 1
Disease progression (General disorders) | 8 | 10
Fatigue (General disorders) | 2 | 0
Multi-organ failure (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1
Abscess (Infections and infestations) | 1 | 0
Fungal skin infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Blood electrolytes abnormal (Investigations) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 4 | 4
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 6
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=25) | Aflibercept (N=30)
Anaemia (Blood and lymphatic system disorders) | 4 | 3
Tachycardia (Cardiac disorders) | 1 | 2
Abdominal distension (Gastrointestinal disorders) | 2 | 5
Abdominal pain (Gastrointestinal disorders) | 5 | 5
Abdominal pain upper (Gastrointestinal disorders) | 1 | 6
Constipation (Gastrointestinal disorders) | 3 | 5
Diarrhoea (Gastrointestinal disorders) | 5 | 12
Dyspepsia (Gastrointestinal disorders) | 2 | 5
Nausea (Gastrointestinal disorders) | 9 | 11
Oral pain (Gastrointestinal disorders) | 0 | 2
Stomatitis (Gastrointestinal disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 13 | 19
Asthenia (General disorders) | 3 | 7
Chest pain (General disorders) | 0 | 2
Fatigue (General disorders) | 14 | 10
Gait disturbance (General disorders) | 1 | 2
Mucosal inflammation (General disorders) | 0 | 2
Oedema peripheral (General disorders) | 10 | 11
Pyrexia (General disorders) | 2 | 3
Nasopharyngitis (Infections and infestations) | 0 | 2
Pneumonia (Infections and infestations) | 0 | 3
Upper respiratory tract infection (Infections and infestations) | 0 | 2
Urinary tract infection (Infections and infestations) | 4 | 1
Weight decreased (Investigations) | 0 | 5
Anorexia (Metabolism and nutrition disorders) | 9 | 8
Dehydration (Metabolism and nutrition disorders) | 2 | 4
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 7
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2
Dizziness (Nervous system disorders) | 1 | 2
Dysgeusia (Nervous system disorders) | 1 | 2
Headache (Nervous system disorders) | 1 | 7
Confusional state (Psychiatric disorders) | 0 | 2
Insomnia (Psychiatric disorders) | 0 | 2
Dysuria (Renal and urinary disorders) | 2 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 3
Proteinuria (Renal and urinary disorders) | 1 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 8
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 6
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 2
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 3
Rash (Skin and subcutaneous tissue disorders) | 2 | 4
Hypertension (Vascular disorders) | 3 | 4
Hypotension (Vascular disorders) | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator shall have the right to independently publish study results from his site after a multicenter publication, or 12 months after the completion of the study by all sites. He must provide the sponsor a copy of any such publication derived from the study for review and comment at least 45 days (20 days) in advance of any submission, and delay publication till the approval of the publication is given in writing by the Sponsor (not to exceed ninety days).